CLINICAL TRIAL: NCT01668368
Title: Goal Directed Mechanical Ventilation Aimed at Optimal Lung Compliance Approach Guided by Esophageal Pressure in Acute Respiratory Failure.
Brief Title: Goal Directed Mechanical Ventilation Aimed at Optimal Lung Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Soroksky Arie, M.D., Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0082-12-WOMC
Record Dates: First submitted 2012-07-23; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Acute Respiratory Failure; ARDS
Keywords: ARDS; Esophageal pressure; pleural pressure; pulmonary compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esophageal balloon group (Other): Esophageal balloon will be inserted, and esophageal pressure will be measured in patients with acute respiratory failure.
  Intervention - PEEP and Inspiratory pressure will be adjusted according to the measured esophageal pressure.
  Interventions: Other: esophageal balloon

INTERVENTIONS:
Other: esophageal balloon — esophageal pressure as a surrogate for pleural pressure
  Other Names: pleural pressure

SUMMARY:
Patients with acute respiratory failure exhibiting decreased respiratory system compliance with hypoxemia or carbon dioxide retention are often difficult to ventilate with current guidelines that limit applied plateau pressure Yet, these guidelines do not take into consideration chest wall mechanics. The investigators sought to determine whether partition of the respiratory system into its components by measuring esophageal pressure and thus assessment of pleural pressure, would help in patients with acute respiratory failure to identify the factors contributing to low respiratory system compliance.

DETAILED DESCRIPTION:
Identifying the dominant factor affecting respiratory system compliance by measuring transpulmonary pressure may better direct and optimize mechanical ventilation. Thus, instead of limiting mechanical ventilation by plateau pressure, PEEP and Inspiratory pressure adjustment would be individualized specifically for each patient's lung compliance as indicated by transpulmonary pressure.

The main goal of this approach is to specifically target transpulmonary pressure instead of plateau pressure, and therefore achieve the best Lung compliance with the least transpulmonary pressure possible.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study a prerequisite of high peak Inspiratory pressure (plateau pressure of up to 30 cmH2O) had to be present, and at least one of the following four inclusion criteria had to be met.

  1 - Low Total Respiratory system compliance (CT), defined as less than 50ml/cmH2O. 2 - P/F ratio of less than 300. 3 - Need for a PEEP greater than 10 cmH2O to maintain SaO2 of > 90%. 4 - PCO2 over 60 mmHg, or PH less than 7.2 that is attributed to respiratory acidosis.

Exclusion Criteria:

* Patients with any of the following were excluded from the study. Previous lung or chest wall surgery, previous esophageal surgery, known Achalasia or any other esophageal motility or spasm disorder, presence of chest thoracostomy tube, and any significant chest wall abnormality such as kyphoskoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Oxygenation | 1 year

SECONDARY OUTCOMES:
lung compliance, expressed as ml/cmH2O. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, MD, Principal Investigator — Wolfson MC

REFERENCES:
- [Result] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507